CLINICAL TRIAL: NCT00770653
Title: Effects of a Pioglitazone/Metformin Fixed Combination in Comparison to Metformin in Combination With Glimepiride on Diabetic Dyslipidemia
Brief Title: Efficacy of Pioglitazone/Metformin Combination Therapy in Subjects With Type 2 Diabetes Mellitus and Dyslipidemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma GmbH, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATS K024; 2006-004455-37 (EudraCT Number); D-PIO-114 (Other: Takeda Pharma GmbH); U1111-1114-1678 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2010-10-06 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus; Dyslipidemias
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Hyperlipidemias; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Hyperlipidemias | interventions — Pioglitazone; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone 15 mg and Metformin 850 mg BID (Experimental)
  Interventions: Drug: Pioglitazone and Metformin
- Glimepiride 2 mg and Metformin 850 mg BID (Active Comparator)
  Interventions: Drug: Glimepiride and Metformin

INTERVENTIONS:
Drug: Pioglitazone and Metformin — Pioglitazone 15 mg/metformin 850 mg combination tablets, orally, twice daily and glimepiride placebo-matching tablets, orally, once daily and metformin placebo-matching tablets, orally, twice daily for up to 24 weeks.
  Other Names: ACTOS®; AD-4833; OPIMET
  Arms: Pioglitazone 15 mg and Metformin 850 mg BID
Drug: Glimepiride and Metformin — Pioglitazone/metformin placebo-matching combination tablets, orally, twice daily and glimepiride 2 mg, tablets, orally, once daily and metformin 850 mg, tablets, orally, twice daily for up to 24 weeks.
  Other Names: Amaryl; Glista
  Arms: Glimepiride 2 mg and Metformin 850 mg BID

SUMMARY:
The purpose of this study is to compare pioglitazone and metformin combination therapy, twice daily (BID), to glimepiride and metformin combination therapy for treating diabetic subjects with dyslipidemia.

DETAILED DESCRIPTION:
Insulin resistance is a major endocrinopathy preceding the development of hyperglycemia, diabetic dyslipidemia and cardiovascular disease in type 2 diabetes. The most common pattern of dyslipidemia in patients with type 2 diabetes are elevated triglyceride levels, decreased hih-density lipoprotein cholesterol and a predominance of small dense low-density lipoprotein particles. Each of these dyslipidemia features is associated with an increased risk of cardiovascular events.

Pioglitazone and Metformin are established drugs which can be used for the treatment of type 2 diabetes. This study will investigate the effects of treatment with fixed Pioglitazone/Metformin combination therapy of Metformin and Glimepiride in Metformin-pretreated type 2 diabetic patients with dyslipidemia.

Total participation time in this study is anticipated to be approximately 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes according to the American Diabetes Association Criteria.
* Treatment with individual maximal tolerated dose of metformin (850 - 2000 mg) as monotherapy within the last 12 weeks.
* Glycosylated Hemoglobin greater than or equal to 6.5% and less than or equal to 9%.
* Dyslipidemia defined as high-density lipoprotein cholesterol less than or equal to 1.03 mmol/l (40 mg/dL) and/or triglycerides greater than or equal to 1.7 mmol/l (150 mg/dL).
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Type 1 diabetes mellitus.
* Insulin-dependent type 2 diabetes mellitus.
* Treatment or history of treatment with any insulin formulation other than emergency for more than 2 weeks.
* Treatment with other oral antidiabetic drugs in addition to metformin within the last 12 weeks.
* Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Heparin (and heparin-like drugs)
  * coumarin
  * phenprocoumon
  * hirudin
  * Protein C
  * Fondaparinux
  * antithrombin III
  * Peroxisome Proliferation Activating Receptor (gamma) agonists
  * Treatment within the last 12 weeks with:

    * fibrates
    * gemfibrozil
    * niacin
    * months
    * Rifampicin
  * Changes in dosage of any statin treatment to lower low-density lipoprotein within 2 weeks before study entry and during study participation interval.
  * Changes in dosage of any anticoagulant treatment with acetyl salicylic acid and/or clopidogrel within 2 weeks before study entry and during study participation interval.
  * Start of statin and/or anticoagulant treatment during study participation interval.
* History of severe or multiple allergies and/ or acute severe infections.
* Have had more than one unexplained episode of severe hypoglycemia (defined as requiring assistance of another person due to disabling hypoglycemia) within 6 months prior to screening visit.
* Progressive fatal disease.
* Any elective surgery during study participation.
* History of drug or alcohol abuse within the last 5 years.
* A history of significant cardiovascular (New York Heart Association stage I - IV), respiratory, gastrointestinal, hepatic (alanine aminotransferase and/or aspartate aminotransferase greater than 2.5 times the upper limit of the normal reference range), renal (serum creatinine greater than 1.2 mg/dL in women and greater than 1.5 mg/dL in men, glomerular filtration rate less than 60 ml/min as estimated by the Cockroft-Gault formula), neurological, psychiatric and/or hematological disease as judged by the investigator, history of macular edema.
* Blood donation within the last 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Adviser Clinical Research, Study Director — Takeda Pharma Gmbh, Aachen (Germany)
Locations (64):
- Germany (64):
  - Bretten, Baden-Wurttemberg
  - Deggingen, Baden-Wurttemberg
  - Dettenheim, Baden-Wurttemberg
  - Künzelsau, Baden-Wurttemberg
  - Rottweil, Baden-Wurttemberg
  - Spaichingen, Baden-Wurttemberg
  - Stockach, Baden-Wurttemberg
  - Wangen, Baden-Wurttemberg
  - Augsburg, Bavaria
  - Feldafing, Bavaria
  - Furth im Wald, Bavaria
  - Immenstadt im Allgäu, Bavaria
  - Lichtenfels, Bavaria
  - München, Bavaria
  - Schweinfurt, Bavaria
  - Waldkraiburg, Bavaria
  - Wallerfing, Bavaria
  - Weilersbach, Bavaria
  - Würzburg, Bavaria
  - Ketzin, Brandenburg
  - Rüdersdorf, Brandenburg
  - Bermerhaven, City state Bremen
  - Hamburg, Hamburg
  - Bensheim, Hesse
  - Ehrenberg, Hesse
  - Gersfeld, Hesse
  - Kassel, Hesse
  - Kelkheim, Hesse
  - Offenbach, Hesse
  - Celle, Lower Saxony
  - Einbeck, Lower Saxony
  - Hanover, Lower Saxony
  - Hildesheim, Lower Saxony
  - Schwerin, Mecklenburg-Vorpommern
  - Bad Berleburg, North Rhine-Westphalia
  - Bad Laasphe, North Rhine-Westphalia
  - Bad Oeynhausen, North Rhine-Westphalia
  - Bocholt, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Dinslaken, North Rhine-Westphalia
  - Dorsten, North Rhine-Westphalia
  - Duisburg, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Frechen, North Rhine-Westphalia
  - Isselburg, North Rhine-Westphalia
  - Kamen, North Rhine-Westphalia
  - Marl, North Rhine-Westphalia
  - Menden, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Siegen, North Rhine-Westphalia
  - Diez, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Neuwied, Rhineland-Palatinate
  - Rodenbach, Rhineland-Palatinate
  - Simmern, Rhineland-Palatinate
  - Borna, Saxony
  - Dresden, Saxony
  - Meissen, Saxony
  - Mittweida, Saxony
  - Magdeburg, Saxony-Anhalt
  - Reinfeld, Schleswig-Holstein
  - Berlin, State of Berlin
  - Altenburg, Thuringia
  - Blankenhain, Thuringia

REFERENCES:
- [Derived] Pfutzner A, Schondorf T, Tschope D, Lobmann R, Merke J, Muller J, Lehmann U, Fuchs W, Forst T. PIOfix-study: effects of pioglitazone/metformin fixed combination in comparison with a combination of metformin with glimepiride on diabetic dyslipidemia. Diabetes Technol Ther. 2011 Jun;13(6):637-43. doi: 10.1089/dia.2010.0233. Epub 2011 Apr 2. PMID 21457065
- See also: ACTOPLUS MET® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOPLUSMETPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 61 investigative sites in Germany from 03 April 2007 to 13 May 2009.
Pre-assignment Details: Subjects with type 2 diabetes with diabetic dyslipidemia, inadequately controlled by Metformin monotherapy were enrolled in one of two, twice-daily (BID) combination therapy treatment groups.
Groups:
- Pioglitazone 15 mg and Metformin 850 mg BID: Pioglitazone 15 mg/metformin 850 mg combination tablets, orally, twice daily and glimepiride placebo-matching tablets, orally, once daily and metformin placebo-matching tablets, orally, twice daily for up to 24 weeks.
- Glimepiride 2 mg and Metformin 850 mg BID: Pioglitazone/metformin placebo-matching combination tablets, orally, twice daily and glimepiride 2 mg, tablets, orally, once daily and metformin 850 mg, tablets, orally, twice daily for up to 24 weeks.
Period: Overall Study
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Started | 155 | 150
Completed | 123 | 121
Not Completed | 32 | 29
Not completed — Adverse Event | 13 | 5
Not completed — Protocol Violation | 8 | 6
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Lack of Compliance | 1 | 4
Not completed — Worsening of Glycosolated Hemoglobin | 2 | 2
Not completed — Fasting Glucose > 240 mg/dL | 2 | 1
Not completed — > Three Moderate Hypoglycemic Episodes | 0 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID | Total
Number analyzed (Participants) | 153 | 149 | 302
Age Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.0) | 58.5 (9.6) | 58.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 99 | 94 | 193
Region of Enrollment [Number; unit: participants]
  Germany | 153 | 149 | 302

OUTCOME MEASURES:

1. Primary Outcome: The Mean Increase From Baseline in High-Density Lipoprotein Cholesterol.
Description: The increase in High-Density Lipoprotein (HDL) Cholesterol collected at week 24 or final visit and HDL-Cholesterol collected at baseline.
Time Frame: Baseline and Week 24.
Population: Analysis was performed on participants with at least one valid baseline and post-baseline measurement. This condition was not fulfilled in 17 participants who were excluded from the all-participants-randomized set, leading to a full-analysis-set of 288 (146 vs. 142). Last observation carried forward was used (LOCF) in case of premature termination.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 146 | 142
mg/dL | 3.2 (9.7) | -0.3 (11.0)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Null hypothesis (H0) = mean increase of HDL after 24 weeks of treatment of Pio/Met group ≤ the mean increase in the Gli/Met group. Alternate hypothesis (H1) = mean increase of HDL after 24 weeks of treatment of Pio/Met group > the mean increase in the Gli/Met group. The relevant clinical effect size to detect with adequate power was 0.35. With this assumption, a one sided t-test with a type I error rate had 80% power to reject the H0 for the H1 when the sample size was 130 patients per group; Test type: Superiority or Other; p = 0.0018, ANCOVA; Mean Difference (Final Values) = 3.2670, 95% CI 2-sided [1.2264 to 5.3076]

2. Secondary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol.
Description: The change between HDL-Cholesterol collected at week 24 or final visit and HDL-Cholesterol collected at baseline.
Time Frame: Baseline and Week 24.
Population: Analyses was performed for the full analysis and per-protocol set. This condition was not fulfilled in some participants who were excluded. Last observation carried forward was used (LOCF) in case of premature termination.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 143 | 137
mg/dL | 3.3 (9.6) | -0.4 (11.1)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0018, ANCOVA; Mean Difference (Final Values) = 3.2670, 95% CI 2-sided [1.2264 to 5.3076] — Deviation from the normal distribution assumption was detected for original and rank-transformed data for all time-points due to p-value of Shapiro-Wilk test, indicating the normal distribution assumption might be distrusted for HDL-cholesterol data

3. Secondary Outcome: Change From Baseline in High-Density Lipoprotein/Low-Density Lipoprotein Ratio.
Description: The change between High-Density Lipoprotein/Low-Density Lipoprotein Ratio collected at week 24 or final visit and High-Density Lipoprotein/Low-Density Lipoprotein Ratio collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 141 | 132
mg/dL | 0.1 (0.8) | 0.3 (0.7)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.1167, ANCOVA; Mean Difference (Final Values) = -0.1311, 95% CI 2-sided [-0.2951 to 0.0329]

4. Secondary Outcome: Change From Baseline in Triglycerides.
Description: The change between the value of Triglycerides collected at week 24 or final visit and Triglycerides collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 146 | 142
mg/dL | -40.9 (113.8) | -16.7 (121.6)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.1012, ANCOVA; Mean Difference (Final Values) = -17.9479, 95% CI 2-sided [-39.4331 to 3.5373]

5. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Subfractions.
Description: The change between the value of Low-Density Lipoprotein Subfractions collected at week 24 or final visit and Low-Density Lipoprotein Subfractions collected at baseline.
Time Frame: Baseline and Week 24.
Population: Analyses was performed for the full analysis and per-protocol set. The number of participants for analysis was derived from a subgroup of participants from the Mainz, Germany study site. Last observation carried forward was used (LOCF) in case of premature termination.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 11
mg/dL | 6.2 (17.5) | 6.1 (26.4)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.7486, ANCOVA; Mean Difference (Final Values) = 3.1292, 95% CI 2-sided [-17.0109 to 23.2693]

6. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol.
Description: The change between Low-Density Lipoprotein Cholesterol collected at week 24 or final visit and Low-Density Lipoprotein Cholesterol collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 143 | 132
mg/dL | 9.7 (34.7) | 11.2 (25.3)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.9464, ANCOVA; Mean Difference (Final Values) = -0.2355, 95% CI 2-sided [-7.1253 to 6.6543]

7. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin.
Description: The change between the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 or final visit and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 139 | 136
mg/dL | -0.83 (0.87) | -0.95 (0.85)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0807, ANCOVA; Mean Difference (Final Values) = 0.1574, 95% CI 2-sided [-0.0193 to 0.3341]

8. Secondary Outcome: Change From Baseline in Fasting Intact Proinsulin.
Description: The change between Fasting Intact Proinsulin collected at week 24 or final visit and Fasting Intact Proinsulin collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 144 | 137
pmol/L | -5.18 (11.89) | -0.11 (9.84)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = -4.5039, 95% CI 2-sided [-6.4222 to -2.5855]

9. Secondary Outcome: Change From Baseline in Fasting Glucose.
Description: The change between Fasting Glucose collected at week 24 or final visit and Fasting Glucose collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 145 | 139
mg/dL | -21.6 (38.6) | -21.1 (40.4)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.7799, ANCOVA; Mean Difference (Final Values) = 1.0707, 95% CI 2-sided [-6.4665 to 8.6079]

10. Secondary Outcome: Change From Baseline in Adiponectin.
Description: The change between Adiponectin collected at week 24 or final visit and Adiponectin collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μg/mL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 146 | 139
μg/mL | 6.79 (6.38) | 0.72 (2.73)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = 6.3161, 95% CI 2-sided [5.0994 to 7.5329]

11. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (Original).
Description: The change between the value of High Sensitivity C-reactive Protein collected at week 24 or final visit and High Sensitivity C-reactive Protein collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 141 | 135
mg/L | -0.21 (8.98) | -0.04 (9.53)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.4131, ANCOVA; Mean Difference (Final Values) = -0.8323, 95% CI 2-sided [-2.8312 to 1.1665]

12. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (≤ 10 mg/L).
Description: The change between the value of High Sensitivity C-reactive Protein less than or equal to 10 mg/L collected at week 24 or final visit and High Sensitivity C-reactive Protein less than or equal to 10 mg/L collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 123 | 113
mg/L | -0.87 (1.88) | 0.00 (1.83)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = -0.8847, 95% CI 2-sided [-1.3067 to -0.4627]

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure.
Description: The change between Systolic Blood Pressure measured at week 24 or final visit and Systolic Blood Pressure measured at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 146 | 142
mmHg | -2.5 (14.8) | 0.5 (13.8)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0929, ANCOVA; Mean Difference (Final Values) = -2.4903, 95% CI 2-sided [-5.3979 to 0.4172]

14. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure.
Description: The change between Diastolic Blood Pressure measured at week 24 or final visit and Diastolic Blood Pressure measured at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 146 | 142
mmHg | -1.3 (8.7) | -0.1 (8.8)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.3279, ANCOVA; Mean Difference (Final Values) = -0.8832, 95% CI 2-sided [-2.6571 to 0.8906]

15. Secondary Outcome: Intake of Study Medication Greater Than 80% and Less Than 120%.
Description: The change between the Intake of study medication greater than 80% at week 24 or final visit and Baseline and the Intake of study medication greater than 80% at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 146 | 142
participants | 136 | 137
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; The number and percentage of participants with a calculated compliance >80% and <120% are presented for both treatment groups. In addition, the p-values of Fisher's exact test, the two-sided 95% confidence intervals for the percentage of patients per treatment group and for the difference between the treatment groups are provided; Test type: Superiority or Other; p = 0.2895, Fisher Exact; Fisher Exact = -3.33, 95% CI 2-sided [-14.83 to 8.39]

16. Secondary Outcome: Change From Baseline in Nitrotyrosine.
Description: The change between the value of Nitrotyrosine collected at week 24 or final visit and Nitrotyrosine collected at baseline.
Time Frame: Baseline and Week 24.
Population: Analyses was performed for the full analysis and per-protocol set. The number of participants for analysis was derived from a subgroup of participants from Schwerin, Berlin, Hanover and Münster study sites. Last observation carried forward was used (LOCF) in case of premature termination.
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 23 | 20
nmol/L | -2.7 (93.2) | 32.5 (147.2)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.3517, ANCOVA; Mean Difference (Final Values) = -29.9516, 95% CI 2-sided [-94.1999 to 34.2967]

17. Secondary Outcome: Change From Baseline in Soluble CD40 Ligand.
Description: The change between the value of Soluble CD40 Ligand collected at week 24 or final visit and Soluble CD40 Ligand collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 16 | 18
pg/mL | -40.7 (248.6) | 102.4 (379.8)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.1979, ANCOVA; Mean Difference (Final Values) = -151.4477, 95% CI 2-sided [-386.2256 to 83.3302]

18. Secondary Outcome: Change From Baseline in Matrix Metallo Proteinase-9.
Description: The change between the value of Baseline in Matrix Metallo Proteinase-9 collected at week 24 or final visit and Baseline in Matrix Metallo Proteinase-9 collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 23 | 20
ng/mL | 31.4 (228.3) | 51.6 (216.4)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.7186, ANCOVA; Mean Difference (Final Values) = -24.8589, 95% CI 2-sided [-163.3229 to 113.6052]

19. Secondary Outcome: Change From Baseline in Soluble Intracellular Adhesion Molecule.
Description: The change between the value of Baseline in Soluble Intracellular Adhesion molecule at week 24 or final visit and Baseline in Soluble Intracellular Adhesion molecule collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 23 | 20
ng/mL | -13.0 (46.9) | -3.2 (50.0)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.5058, ANCOVA; Mean Difference (Final Values) = -9.9728, 95% CI 2-sided [-39.9915 to 20.0459]

20. Secondary Outcome: Change From Baseline in Soluble Vascular Cell Adhesion Molecule.
Description: The change between the value of Soluble Vascular Cell Adhesion Molecule collected at week 24 or final visit and Soluble Vascular Cell Adhesion Molecule collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 22 | 20
ng/mL | 11.6 (160.6) | 3.3 (115.4)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.5230, ANCOVA; Mean Difference (Final Values) = 28.3988, 95% CI 2-sided [-60.7193 to 117.5169]

21. Secondary Outcome: Change From Baseline in Thromboxane B2.
Description: The change between the value of Thromboxane B2 collected at week 24 or final visit and Thromboxane B2 collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 19 | 20
pg/mL | -216.4 (842.9) | 527.8 (1190.4)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.2203, ANCOVA; Mean Difference (Final Values) = -367.2639, 95% CI 2-sided [-964.3923 to 229.8646]

22. Secondary Outcome: Change From Baseline in Platelet Function.
Description: The change between the value of Platelet Function by PFA 100 collected at week 24 or final visit and Platelet Function by PFA 100 collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: sec
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 3 | 5
sec | -30.3 (44.3) | -1.0 (102.5)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.5850, ANCOVA; Mean Difference (Final Values) = 28.0794, 95% CI 2-sided [-95.6468 to 151.8057]

23. Secondary Outcome: Change From Baseline in E-Selectin.
Description: The change between the value of E-Selectin collected at week 24 or final visit and E-Selectin collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 23 | 20
ng/mL | -3.7 (4.8) | -0.5 (3.4)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0138, ANCOVA; Mean Difference (Final Values) = -2.4205, 95% CI 2-sided [-4.3207 to -0.5202]

24. Secondary Outcome: Change From Baseline in Von-Willebrand Factor.
Description: The change between the value of Von-Willebrand Factor collected at week 24 or final visit and Von-Willebrand Factor collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 24 | 20
percent | -19.5 (32.0) | 1.4 (33.2)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0817, ANCOVA; Mean Difference (Final Values) = 0.0009, 95% CI 2-sided [-30.1139 to 1.8578]

25. Secondary Outcome: Change From Baseline in Erythrocyte Deformability (0.30%).
Description: The change between the 0.30 percent value of Erythrocyte (Red Blood Cell) Deformability collected at week 24 or final visit and Erythrocyte Deformability collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 12
percent | 1.3 (2.1) | -0.4 (1.7)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.1761, ANCOVA; Mean Difference (Final Values) = 0.9935, 95% CI 2-sided [-0.4843 to 2.4712]

26. Secondary Outcome: Change From Baseline in Erythrocyte Deformability (0.60%)
Description: The change between the 0.60 percent value of Erythrocyte (Red Blood Cell) Deformability collected at week 24 or final visit and Erythrocyte Deformability collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 12
percent | 2.4 (1.3) | -0.5 (1.1)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = 2.5263, 95% CI 2-sided [1.3832 to 3.6695]

27. Secondary Outcome: Change From Baseline in Erythrocyte Deformability (1.20).
Description: The change between the 1.20 percent value of Erythrocyte (Red Blood Cell) Deformability collected at week 24 or final visit and Erythrocyte Deformability collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 12
percent | 3.2 (2.2) | -1.1 (2.5)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0055, ANCOVA; Mean Difference (Final Values) = 3.2345, 95% CI 2-sided [1.0675 to 5.4016]

28. Secondary Outcome: Change From Baseline in Erythrocyte Deformability (3.00).
Description: The change between the 3.00 percent value of Erythrocyte (Red Blood Cell) Deformability collected at week 24 or final visit and Erythrocyte Deformability collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 12
percent | 3.3 (2.8) | -.15 (3.1)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0264, ANCOVA; Mean Difference (Final Values) = 2.9712, 95% CI 2-sided [0.3863 to 5.5562]

29. Secondary Outcome: Change From Baseline in Erythrocyte Deformability (6.00).
Description: The change between the 6.00 percent value of Erythrocyte (Red Blood Cell) Deformability collected at week 24 or final visit and Erythrocyte Deformability collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 12
percent | 3.1 (2.9) | -1.4 (2.9)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.0509, ANCOVA; Mean Difference (Final Values) = 2.5394, 95% CI 2-sided [-0.0114 to 5.0901]

30. Secondary Outcome: Change From Baseline in Erythrocyte Deformability (12.00).
Description: The change between the 12.00 percent value of Erythrocyte (Red Blood Cell) Deformability collected at week 24 or final visit and Erythrocyte Deformability collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 12
percent | 2.7 (2.8) | -1.3 (2.9)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.1013, ANCOVA; Mean Difference (Final Values) = 2.1718, 95% CI 2-sided [-0.4660 to 4.8097]

31. Secondary Outcome: Change From Baseline in Erythrocyte Deformability (30.00).
Description: The change between the 30.00 percent value of Erythrocyte (Red Blood Cell) Deformability collected at week 24 or final visit and Erythrocyte Deformability collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 12
percent | 2.5 (2.6) | -1.3 (3.5)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.1363, ANCOVA; Mean Difference (Final Values) = 2.1346, 95% CI 2-sided [-0.7338 to 5.0031]

32. Secondary Outcome: Change From Baseline in Erythrocyte Deformability (60.00).
Description: The change between the 60.00 percent value of Erythrocyte (Red Blood Cell) Deformability collected at week 24 or final visit and Erythrocyte Deformability collected at baseline.
Time Frame: Baseline and Week 24.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Number analyzed (Participants) | 11 | 12
percent | 2.7 (2.6) | -1.3 (3.9)
Statistical Analysis 1: Comparison: Pioglitazone 15 mg and Metformin 850 mg BID vs Glimepiride 2 mg and Metformin 850 mg BID; Test type: Superiority or Other; p = 0.1165, ANCOVA; Mean Difference (Final Values) = 2.4181, 95% CI 2-sided [-0.6561 to 5.4922]

ADVERSE EVENTS:
Time Frame: 1 year and 11 months. Treatment-emergent adverse events are defined as those occurring after signature of consent form and no more than 14 days after the end of the study.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Irrespective of the relation to study treatment, any event spontaneously reported by the participant or observed by the investigator was recorded.
Arm/Group | Pioglitazone 15 mg and Metformin 850 mg BID | Glimepiride 2 mg and Metformin 850 mg BID
Serious Adverse Events (participants affected / at risk) | 17/153 | 8/149
Other Adverse Events (participants affected / at risk) | 61/153 | 61/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone 15 mg and Metformin 850 mg BID (N=153) | Glimepiride 2 mg and Metformin 850 mg BID (N=149)
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Tumour marker increased (Investigations) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone 15 mg and Metformin 850 mg BID (N=153) | Glimepiride 2 mg and Metformin 850 mg BID (N=149)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 14 | 14
Headache (Nervous system disorders) | 7 | 7
Nasopharyngitis (Infections and infestations) | 24 | 33
Oedema peripheral (General disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 14 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.